CLINICAL TRIAL: NCT01129908
Title: Saliva Composition and Oral Hygiene in Children With Celiac Disease Before and After the Change in Diet
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Moti Moskovitz, Clinical Senior Lecturer, Hadassah Medical Organization
Other Study IDs: odelia- HMO-CTIL
Record Dates: First submitted 2010-05-23; First posted 2010-05-25 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Celiac Disease
Keywords: oral health in children with celiac disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The celiac disease (CD) is a disease with an immune and genetic component that is activated by the presence of gluten, and damages the intestine mucosa and causes malabsorption of food.

In the oral environment the investigators see enamel defects and recurrent ulcers.

Celiac patients have to keep a restrict gluten-free diet, in order to prevent the clinical symptoms of the disease (such as diarrhea, stomach ache and weight loss).

It has been assumed that the patients have less cariogenic diet, and that caries prevalence is not as high as in normal population.

In celiac patients the investigators find enamel defects that are characterized with pits and deep fissures and sometimes the complete loss of enamel. These defects are classified by the grading of the CD related DED's (dental enamel defects) according to Aine. These defects are symmetrical defects in the permanent dentition, in teeth that develops at the same time. The cause is thought to be hypocalcaemia or genetic.

These defects were found in 42.2% of celiac patients in appose to only 5.4% in healthy population.

Recurrent ulcers were found in 41% in the oral cavity of celiac patients, compare to 27% in healthy population.

After changing the diet to a gluten-free diet, an improvement is seen in the presence of these ulcers.

ELIGIBILITY:
Inclusion Criteria:

* celiac disease

Exclusion Criteria:

* no other systemic condition
* age 3-18
* children on medication

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: chilren with celiac disease
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)